CLINICAL TRIAL: NCT00635856
Title: Phase II, Open-Label Trial to Assess the Activity of ZD1839 (IRESSA TM) in Patients With Recurrent Prostate Cancer Who Have Rising Serum PSA Levels Despite Serum Testosterone < 50mg/dl
Brief Title: Open Label Trial to Assess Iressa in Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Alison Armour Medical Science Director, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1839US/0040; NCT00033579 (obsolete NCT alias)
Expanded Access: Available
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Prostate Cancer
Keywords: Iressa; Gefitinib; Prostate Cancer; PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gefitinib — Iressa

SUMMARY:
A study to assess the activity of Iressa in patients who's prostate cancer has recurred, and who have rising PSA levels

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer diagnosis
* no evidence of metastasis
* Age 18 or older

Exclusion Criteria:

* Prior chemotherapy for recurrent prostate cancer
* Radiotherapy completed within 28 days of starting the study
* Incomplete healing from prior cancer or other major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2001-05; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Serum Prostate Specific Antigen | Monthly

SECONDARY OUTCOMES:
Duration of PSA decline | Monthly
Safety variables | Monthly
Time to Progression | Every 3 months